CLINICAL TRIAL: NCT02087410
Title: Ghrelin in Polycystic Ovary Syndrome
Brief Title: Serum Ghrelin in Polycystic Ovary Syndrome
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: amr hesham el etreby (Other)
Responsible Party: Sponsor-Investigator, amr hesham el etreby, resident maternity hospital, Ain Shams University
Organization: Ain Shams University (Other)
Other Study IDs: Ghrelin
Record Dates: First submitted 2014-03-12; First posted 2014-03-14 (Estimated); Last update posted 2014-03-14 (Estimated); Status verified 2014-03

CONDITIONS: Polycystic Ovary
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — blood sample
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- study: patients with polycystic ovary syndrome
- control: healthy patients serves as control group

SUMMARY:
measuring serum gherlin in polycystic ovary syndrome patients and compare it to healthy levels

DETAILED DESCRIPTION:
two groups one healthy and other with pco measure ghrelin level in both of them to find relation between pco and ghrelin

ELIGIBILITY:
Inclusion Criteria:pco women

* At least 12 months of infertility.
* Patients with polycystic ovarian syndrome according to Rotterdam criteria:

Exclusion Criteria:

* Patients with hyperprolactinemia
* Patients with Cushing's syndrome
* Patients with Congenital or non-classical adrenal hyperplasia
* Patients with hormone secreting tumors.
* Patients with hormonal treatment in the last 3 months.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Forty two patients with polycystic ovarian syndrome and forty two healthy subjects will be recruited from the outpatient clinic Ain Shams University Maternity Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2014-04; Primary Completion 2014-10 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
relationships between circulating ghrelin and the clinical and biochemical manifestations of PCOS | after 6 monthes
  Analysis of levels of ghrelin in study group

CONTACTS AND LOCATIONS:
Overall Officials: amr eletrby, MBBCH, Principal Investigator — ain shams universty maternity hospital
Locations (1):
- Maternity Hospital, Cairo, Cairo Governorate, Egypt